CLINICAL TRIAL: NCT02534012
Title: Paravertebral Block Versus General Anesthesia for Major Abdominal Surgery in Elderly: a Prospective Randomized Clinical Trial
Brief Title: Paravertebral Block vs. General Anesthesia for Major Abdominal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Zoher Naja, Chairperson of Anesthesia and Pain Management Department, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 182015
Record Dates: First submitted 2015-08-20; First posted 2015-08-27 (Estimated); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Major Abdominal Surgery
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PVB group (Experimental): Patients will receive nerve stimulator guided paravertebral block
  Interventions: Drug: Paravertebral block; Procedure: Major abdominal surgery
- GA group (Experimental): Patients will receive general anesthesia
  Interventions: Drug: General anesthesia; Procedure: Major abdominal surgery

INTERVENTIONS:
Drug: Paravertebral block — Bilateral nerve stimulator-guided PVB is performed while patients are in lateral decubitis position. An intervertebral line is drawn at the appropriate levels and the injection site is marked 2.5 cm lateral to the midline on both sides. After aseptic preparation of the skin, 0.3 mL 2% lidocaine is infiltrated at the injection sites. A 22-G nerve stimulation needle (Stimuplex, B.Braun, Melsungen, Germany) is advanced 1-2 cm perpendicularly to the skin using a nerve stimulating current of 2.5-5.0 mA, while closely watching for contractions of the abdominal muscles. The tip of the needle is adjusted to continue to produce muscle contractions while reducing the stimulating current to approximately 0.5-0.6 mA. Depending on patient weight, 3-5 mL of the local anaesthetic mixture is injected at each injection site.
  Arms: PVB group
Drug: General anesthesia — Anesthesia is induced with 1 µg/kg fentanyl, 1.5-2 mg/kg propofol and 1-2 mg midazolam. Then, endotracheal intubation is facilitated by 0.15 mg nimbex (cisatracurium). Anesthesia is maintained by 1-1.5% sevoflurane, 0.5 µg/kg/h fentanyl, 0.05 mg/kg/h nimbex, 60% nitrous oxide and 40% oxygen.
  Arms: GA group
Procedure: Major abdominal surgery

SUMMARY:
Elderly patients are usually presented with higher risk for developing cardiopulmonary complications after general anesthesia (GA). Bilateral paravertebral block (PVB) has been associated with favorable outcomes in patients undergoing ventral hernia repair. Hence, elderly patients undergoing major abdominal surgery may benefit from PVB anesthetic technique.

DETAILED DESCRIPTION:
Introduction

Elderly patients are usually presented with higher risk for developing cardiopulmonary complications after general anesthesia (GA). The risk of adverse events in elderly patients increases with the combination of intraoperative fentanyl, opioid premedication and neuromuscular blockers. Bilateral paravertebral block (PVB) has been associated with favorable outcomes in patients undergoing ventral hernia repair. Hence, elderly patients may benefit from PVB anesthetic technique.

The objective of the study is to compare PVB versus GA for elderly patients undergoing major abdominal surgery. The primary outcome measure is admission to the Intensive Care Unit (ICU). The secondary objective is postoperative analgesic consumption.

Methods

Following approval from the Institutional Review Board, 60 patients aged 70 years or older scheduled to undergo major abdominal surgery from May 2016 till December 2020 will be included in the study. Consent will be obtained from the patients or their family member. Patients will be divided into two groups. Group I will receive PVB while group II will receive GA.

Demographic variables including age, gender, height, weight, and ASA physical status will be collected for each patient. Intraoperative hemodynamic data such as mean arterial pressure (MAP) and heart rate (HR) are noted. Moreover, surgery duration, admission to ICU and hospital stay are recorded. Morbidity and mortality rates will also be obtained.

General Anesthesia technique Anesthesia is induced with 1 µg/kg fentanyl, 1.5-2 mg/kg propofol and 1-2 mg midazolam. Then, endotracheal intubation is facilitated by 0.15 mg nimbex. Anesthesia is maintained by 1-1.5% sevoflurane, 0.5 µg/kg/h fentanyl, 0.05 mg/kg/h nimbex, 60% nitrous oxide and 40% oxygen. Any hemodynamic change of 25% results in a gradual increase or decrease of the sevoflurane concentration.

Paravertebral Block Technique Bilateral nerve stimulator-guided PVB is performed while patients are in lateral decubitis position. The number and level of injections depend on the type of surgery and length of incision.

The appropriate levels for the PVBs are determined by palpation of the spinous processes. An intervertebral line is drawn at the appropriate levels and the injection site is marked 2.5 cm lateral to the midline on both sides. After aseptic preparation of the skin, 0.3 mL 2% lidocaine is infiltrated at the injection sites. A 22-G nerve stimulation needle (Stimuplex; B. Braun, Melsungen, Germany) is advanced 1-2 cm perpendicularly to the skin using a nerve stimulating current of 2.5-5.0 mA, while closely watching for contractions of the abdominal muscles. The tip of the needle is adjusted to continue to produce muscle contractions while reducing the stimulating current to approximately 0.5-0.6 mA.

Depending on patient weight, 3-5 mL of the local anaesthetic mixture is injected at each injection site. Each 20 mL of the local anaesthetic mixture contains: 8mL lidocaine 2%, 8 mL lidocaine 2% with epinephrine 5µg mL-1, and 4 mL bupivacaine 0.5%.

In case of PVB failure, patients will be converted to GA.

Admission to ICU and hospital stay Patients who are hemodynamically stable, conscious and do not feel pain will be transferred from the PACU to the floor. On the other hand, patients will be admitted to ICU if they are unconscious, intubated, and hemodynamically unstable. Patients will be discharged from hospital when they are able to drink, eat and do not have complications.

Morbidity and complications Morbidity is defined as having chest infection, kidney failure, myocardial infarction, and dementia.

ELIGIBILITY:
Inclusion Criteria:

* Age 70 years or older admitted for major abdominal surgery

Exclusion Criteria:

* Known history of allergic reactions to local anesthesia
* Neurological disorders
* Bleeding disorders
* Infection at site of injection.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-05-01 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Number of patients admitted to Intensive Care Unit (ICU) | 48 hours postoperatively

SECONDARY OUTCOMES:
Hemodynamic stability measured through Mean Arterial Pressure (mmHg) | 48 hours postoperatively
Hemodynamic stability measured through heart rate (beats per minute) | 48 hours postoperatively

OTHER OUTCOMES:
Number of patients who passed away | 48 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Zoher Naja, MD, Principal Investigator — Makassed General Hospital
Locations (1):
- Makassed General Hospital, Beirut, Lebanon